CLINICAL TRIAL: NCT06918132
Title: Phase II Single Arm Study of Neoadjuvant Dual Checkpoint Blockade With Programmed Death-ligand 1 (PD1) and Lymphocyte Activation Gene 3 (LAG-3) Inhibition in Resectable Non-Small Cell Lung Cancer (N-PLANC)
Brief Title: Cemiplimab and Fianlimab Before Surgery for the Treatment of Stage IB-IIIB Non-Small Cell Lung Cancer
Acronym: N-PLANC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230202; NCI-2025-02153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-011212 (Other: Mayo Clinic Institutional Review Board); MC230202 (Other: Mayo Clinic)
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cemiplimab, fianlimab) (Experimental): Patients receive cemiplimab IV over 30 minutes on day 1 of each cycle and fianlimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI during screening, tissue sample collection on study and blood sample collection on study and follow-up. Patients may undergo SOC surgery post-treatment.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Biological: Fianlimab; Procedure: Magnetic Resonance Imaging; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
Biological: Fianlimab — Given IV
  Other Names: Anti-LAG-3 MoAb REGN3767; REGN 3767; REGN3767; WHO 11182
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Surgical Procedure — Undergo SOC surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, Not Otherwise Specified (NOS); Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial tests how well a fixed dose combination (FDC) of cemiplimab and fianlimab before surgery (neoadjuvant) works in treating patients with stage IB-IIIB non-small cell lung cancer (NSCLC). The current standard of care (SOC) for NSCLC is to give chemotherapy and immunotherapy before going to surgery to have the cancer removed (neoadjuvant therapy). Immunotherapy with monoclonal antibodies, such as cemiplimab and fianlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving a FDC of cemiplimab and fianlimab before surgery may kill more tumor cells in treating patients with stage IB-IIIB NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess efficacy of neoadjuvant cemiplimab and fianlimab in patients with resectable/early-stage NSCLC with programmed death-ligand 1 (PD-L1) 1-49%, as measured by rate of major pathologic response (MPR) (defined as ≤ 10% viable tumor cells in resected tumor and lymph nodes).

II. To assess efficacy of neoadjuvant cemiplimab and fianlimab in patients with resectable/early-stage NSCLC with PD-L1 ≥ 50%, as measured by rate of major pathologic response (MPR).

SECONDARY OBJECTIVES:

I. Assess the following endpoints (overall and by PD-L1 subsets): event-free survival (EFS), overall survival (OS), disease-free survival (DFS), response rate, pathological complete response rate (pCR), surgical feasibility, and adverse events.

OTHER GOALS (done overall and by PD-L1 subsets):

I. Assess the following in an exploratory fashion: residual viable tumor cells using various cutpoints, whole exome sequencing (WES), gene copy number analysis, circulating tumor deoxyribonucleic acid (DNA) (ctDNA) analysis, tumor microenvironment (TME) analysis, microbiome analyses, temporal biomarker changes.

II. Assess LAG-3 expression on immune-cells by immunohistochemistry (IHC) (17B4) and major histocompatibility complex class II (MHC-II) and fibrinogen-like protein 1 (FGL1) expression by on tumor cells and correlate with clinical data like MPR rate, EFS, and OS.

III. Determine any correlation between the above biomarkers with clinical data of interest like the MPR rate, EFS, and OS.

IV. Determine ctDNA testing as a marker for minimal residual disease (MRD) and molecular recurrence.

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1 of each cycle and fianlimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) during screening, tissue sample collection on study and blood sample collection on study and follow-up. Patients may undergo SOC surgery post-treatment.

After completion of study treatment, patients are followed up at 90 days, then every 3 months post-surgery for the first 2 years, then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Disease characteristics:

  * Histologically or cytologically confirmed stage IB-IIIB (N2) non-small cell lung cancer (NSCLC) per American Joint Committee on Cancer (AJCC) Cancer Staging Manual Eighth Edition
  * T4 tumors will only be eligible if they are defined as T4 based only on their size (more than 7 cm). All other T4 tumors will be ineligible.
  * Pathologic status of lymph nodes must be known
  * PD-L1 expression ≥ 1% by tumor proportion score (TPS) using immunohistochemistry (IHC)

    * Group A: PD-L1 expression ≥ 1% < 50%
    * Group B: PD-L1 expression ≥ 50%
  * Complete surgical resection of the primary NSCLC must be deemed achievable by thoracic surgeon at screening
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate pulmonary function ascertained by treating surgeon obtained ≤ 30 days prior to registration. A pre- or post-bronchodilator forced expiratory volume in 1 second (FEV1) of 1.0 L and > 40% postoperative predicted value and diffusing capacity of the lungs for carbon monoxide (DLCO) > 40% predicted value are required prior to enrollment
* Hemoglobin ≥ 8.0 g/dL (obtained ≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 15 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (obtained ≤ 15 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained ≤ 15 days prior to registration)
* Calculated creatinine clearance ≥ 45 ml/min using the Chronic Kidney Disease Epidemiology (CKD-EPI) Creatinine Equation (obtained ≤ 15 days prior to registration)
* Negative pregnancy test done ≤ 8 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ highly effective contraception during the study and up to 6 months after the last dose
* Presence of targetable alterations [Epiderman Growth Factor Receptor (EGFR), anaplastic lymphoma kinase (ALK), receptor tyrosine kinase (ROS1)] in tumor
* Unresectable or metastatic disease
* Active or history of the following:

  * Prior systemic anti-cancer therapy or radiation therapy for the same cancer being studied in this protocol
  * Interstitial lung disease (e.g., idiopathic pulmonary fibrosis or organizing pneumonia), or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or pneumonitis within the last 5 years
  * Autoimmune disease (including any history of inflammatory bowel disease)
  * Any syndrome that required systemic steroids or immunosuppressive medications EXCEPTIONS: patients with vitiligo; resolved childhood asthma/atopy; residual hypothyroidism that requires only hormone replacement; or psoriasis not requiring systemic treatment, type-1 diabetes mellitus, or rheumatoid arthritis managed without disease modifying anti-rheumatic drugs or >10 mg prednisone equivalent
* Patients requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications ≤14 days prior to registration.

NOTE: Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease

* Patients with organ transplantation
* History of myocardial infarction ≤ 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias; or prior immune-related myocarditis
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Uncontrolled infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) or diagnosis of immunodeficiency that is related to, or results in chronic infection.

Note: No testing is required for this study unless mandated by local health authority.

EXCEPTIONS:

* Patients with known HIV who have controlled infection [undetectable viral load and cluster of differentiation 4 (CD4) count above 350 either spontaneously or on a stable antiviral regimen] are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
* Patients with known hepatitis B (hepatitis B surface antigen positive [HBsAg+]) who have controlled infection (serum hepatitis B virus DNA polymerase chain reaction (PCR) that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
* Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV ribonucleic acid (RNA) by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
* Patients with HIV or hepatitis must be reviewed by a qualified specialist (e.g., infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial

  * Receiving any other investigational agent which would be considered as a treatment for the primary malignancy
  * Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
  * Prior malignancy active ≤ 3 years prior to registration except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast, or papillary thyroid
  * Known hypersensitivity to the active substances or to any of the excipients
  * Receipt of live vaccine ≤ 30 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) rate (Group A) | Up to 2 years
  Will be defined as ≤ 10% viable tumor cells in resected tumor and lymph nodes. Will be conducted using two parallel Simon two-stage trial designs. Will be evaluated within the PD-L1 1-49% group.
MPR rate (Group B) | Up to 2 years
  Will be defined as ≤ 10% viable tumor cells in resected tumor and lymph nodes. Will be conducted using two parallel Simon two-stage trial designs. Will be evaluated within the PD-L1 ≥ 50% group.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 5 years
  Defined as the time from study entry to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause (whichever occurs first).
Overall survival (OS) | Up to 5 years
  Defined as the time from study entry to death from any cause.
Disease-free survival (DFS) | Up to 5 years
  Defined as the time from surgery to the first of either disease recurrence or death from any cause.
Overall response rate (ORR) | Up to 5 years
  Will be calculated based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. A tumor response is defined to be either a complete response or partial response noted as the objective status during neoadjuvant treatment.
Pathologic complete response (pCR) rate | Up to 5 years
  Defined as 0% residual viable tumor (complete absence of tumor) in the resected lung and lymph node tissue. Will be reported as pCR rate, defined as the proportion of patients who achieve pCR after neoadjuvant treatment at the time of resection
Surgical feasibility - to surgery | Up to 5 years
  Will be assessed by the number of participants who make it to surgery
Surgical feasibility - complete surgery | Up to 5 years
  Will be assessed by the number of participants who complete surgery
Incidence of adverse events | Up to 90 days after last study treatment, up to 2 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Frequency and percentage of Grade 3+ adverse events will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal Parikh, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials